CLINICAL TRIAL: NCT01348360
Title: Evaluation of Effectiveness and Safety of NOBORI Stent in Routine Clinical Practice; A Multicenter, Prospective, Observational Study
Brief Title: Evaluation of Effectiveness and Safety of NOBORI Stent
Acronym: IRIS-NOBORI
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Terumo Corporation (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD, PhD, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Other Study IDs: CVRF2010-02
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NOBORI stent

SUMMARY:
The objective of this study is to evaluate effectiveness and safety of Nobori stent in the "real world" daily practice as compared with first-generation drug-eluting stents (sirolimus- or paclitaxel-eluting stents).

DETAILED DESCRIPTION:
This study is a non-randomized, prospective, open-label registry to compare the efficacy and safety of NOBORI stents versus first-generation DES in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving NOBORI stents.
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site.

Exclusion Criteria:

* Patients with a mixture of other DESs.
* Terminal illness with life expectancy <1 year.
* Patients with cardiogenic shock.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with coronary artery disease requiring drug eluting stents
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
composite of death, nonfatal myocardial infarction (MI), or ischemic-driven Target- Vessel Revascularization (TVR) | 12 months post procedure

SECONDARY OUTCOMES:
Death (all cause and cardiac) | one month
Death (all cause and cardiac) | 6 months
Death (all cause and cardiac) | yearly up to 5 years
MI | one month
MI | 6 months
MI | yearly up to 5 years
Composite of death or MI | one month
Composite of cardiac death or MI | one month
Composite of cardiac death or MI | 6 months
Composite of cardiac death or MI | yearly and up to 5 years
Composite of death or MI | 6 months
Composite of death or MI | yearly up to 5 years
TVR | one month
TVR | 6 months
TVR | yearly up to 5 years
Target-lesion revascularization (TLR) | one month
Target-lesion revascularization (TLR) | 6 months
Target-lesion revascularization (TLR) | yearly up to 5 years
Stent thrombosis (ARC criteria) | one month
Stent thrombosis (ARC criteria) | 6 months
Stent thrombosis (ARC criteria) | yearly up to 5 years
Procedural success (defined as achievement of a final diameter stenosis of <30% by visual estimation, without the occurrence of death, Q-wave MI, or urgent revascularization during the index hospitalization) | At discharge from the index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center; Ki Bae Seung, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital, Catholic University of Korea
Locations (26):
- South Korea (26):
  - Asan Medical Center, Seoul, Republic of Korea
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - The Catholic University of Korea, Bucheon ST.Mary's Hospital, Bucheon-si
  - Gangwon National Univ. Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Asan Medical Center, Gangneung
  - Chonnam National University Hospital, Gwangju
  - DongGuk University Gyongju Hospital, Gyeongju
  - National Health Insurance Corporation Ilsan Hospital, Ilsan
  - Gachon University Gil Hospital, Incheon
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Kwangju Christian Hospital, Kwangju
  - KangBuk Samsung Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Korea University Hospital, Seoul
  - Kyung Hee University Medical Hospital, Seoul
  - St. Mary's Catholic Medical Center, Seoul
  - The Catholic University of Korea St.Paul's Hospital, Seoul
  - The Catholic University of Korea Yeouido St.Mary's Hospital, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
  - The Catholic University of Korea Uijeongbu St. Mary's Hospital, Uijeongbu-si
  - Ulsan University Hospital, Ulsan